CLINICAL TRIAL: NCT04442633
Title: Clinical Evaluation of Glutamine Combined With Topical Corticosteroids in the Treatment of Erosive Oral Lichen Planus
Brief Title: Glutamine With Topical Corticosteroids for Lichen Planus Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Glutamine and lichen planus
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Lichen Penis Planus
MeSH Terms: interventions — Triamcinolone; Orabase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional therapy (Active Comparator): topical corticosteroid plus antifungal
  Interventions: Drug: Miconazole Oral gel; Drug: Kenacort in orabase
- Glutamine with a topical corticosteroid plus antifungal (Experimental): Glutamine therapy in combination with a topical corticosteroid plus antifungal
  Interventions: Drug: Glutamine Cap/Tab; Drug: Miconazole Oral gel; Drug: Kenacort in orabase

INTERVENTIONS:
Drug: Glutamine Cap/Tab — Glutamine Capsules: One capsule three times daily on an empty stomach for one month
  Arms: Glutamine with a topical corticosteroid plus antifungal
Drug: Miconazole Oral gel — Miconazole oral gel: applied three to four times daily for three weeks
Drug: Kenacort in orabase — Kenacort in orabase: applied two to three times a day for 3 weeks followed by tapering the following 9 weeks until a maintenance dose of two to three times a week is reached

SUMMARY:
Lichen planus (LP) is an inflammatory skin disease of unknown etiology. Glutamine promotes protein and collagen synthesis, imparts immunity, and maintains the alimentary canal mucosa structure.

DETAILED DESCRIPTION:
Lichen planus (LP) is an inflammatory skin disease of unknown etiology. Recently, increased oxidative stress has been implicated in the pathogenesis of erosive oral lichen planus (EOLP). Glutamine is a source of energy for fibroblasts, immunocompetent cells, and intestinal epithelial cells involved in collagen production. It promotes protein and collagen synthesis, imparts immunity, and maintains the alimentary canal mucosa structure.

The aim of this study is to evaluate the effect of Glutamine combined with topical corticosteroid in the treatment of oral erosive LP.

Thirty patients with a confirmed clinical and histopathologic diagnosis of OLP recruited in this study and divided into 2 equal groups, each consisting of 15 subjects. Group 1 consists of patients treated with topical steroids plus antifungal (conventional therapy); Group 2 consists of patients treated with Glutamine combined with topical steroids plus antifungal.

ELIGIBILITY:
Inclusion Criteria:

1. Patients clinically and histopathologically diagnosed to be suffering from EOLP.
2. Patients who had symptoms i.e. pain and/or burning sensation secondary to EOLP.
3. Patients under stressful life conditions as evidenced by ISMA-UK Stress Questionnaire
4. Males and Females with an age ranging from 30-60years

Exclusion Criteria:

1. Patients suspected to have a lichenoid drug reaction or lichenoid contact allergy.
2. Patients suffering from any systemic diseases (such as diabetes, cardiovascular, liver disorder, renal dysfunction)
3. Patients with findings of any physical or mental abnormality which would interfere with or be affected by the study procedure.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Change in oral lichen planus lesions severity | at baseline, 1 months and 3 months
  Mucosal lesion severity score 0: no lesion score 1: white lesion score 2:atrophy/erosion intermixed or not with white lesion score 3: ulceration intermixed or not with white lesion

SECONDARY OUTCOMES:
Change in pain level | at baseline, 1 months and 3 months
  Pain score score 0= no pain score 1= mild score 2= moderate score 3= severe

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral medicine Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Egypt